CLINICAL TRIAL: NCT07057648
Title: Shape-sensing Robotic-assisted Bronchoscopy (ssRAB) for Diagnosis of Peripheral Pulmonary Nodules: A Prospective Cohort Study in Korea
Brief Title: Shape-Sensing Robotic-Assisted Bronchoscopy for Diagnosis of Peripheral Pulmonary Nodules in Korea
Acronym: ssRAB
Status: Not yet recruiting | Type: Observational
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-06-002
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Lung Nodules; Peripheral Lung Lesions; Pulmonary Nodules; Lung Cancers; Bronchoscopy
Keywords: Shape-sensing robotic-assisted bronchoscopy; ssRAB; Robotic bronchoscopy; Peripheral lung nodules; Diagnostic yield; Lung Nodules; Navigation bronchoscopy; Lung biopsy; Korea; Prospective cohort
MeSH Terms: conditions — Multiple Pulmonary Nodules; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ssRAB Cohort: Patients with peripheral lung nodules who undergo shape-sensing robotic-assisted bronchoscopy (ssRAB) for tissue sampling and diagnosis. All participants receive the same procedure using the ION endoluminal system to navigate to peripheral lung nodules and obtain tissue samples for histological diagnosis.
  Interventions: Device: Shape-sensing Robotic-assisted Bronchoscopy (ssRAB)

INTERVENTIONS:
Device: Shape-sensing Robotic-assisted Bronchoscopy (ssRAB) — Diagnostic procedure using the ION endoluminal system (Intuitive Surgical, Sunnyvale, CA) for navigation and tissue sampling of peripheral pulmonary nodules. The procedure involves:
  1. Pre-procedure 3D navigation planning using thin-section chest CT
  2. Shape-sensing catheter navigation to target nodules
  3. Real-time position monitoring with fiber optic sensors
  4. Tissue sampling using various tools (biopsy needles, forceps, brush, or cryobiopsy)
  5. Optional radial endobronchial ultrasound (rEBUS) confirmation
  6. Fluoroscopic guidance when needed
  The procedure is performed under deep sedation or general anesthesia through an endotracheal tube.

SUMMARY:
What is this study about? This study tests a new robotic technology to take tissue samples from lung nodules (small spots in the lungs). Some lung nodules are cancer, but doctors need a tissue sample to know for sure.

What is the problem? Current methods to get tissue from lung nodules only work about 7 out of 10 times. When they don't work, doctors may need riskier procedures.

What is the new technology? The new technology is called robotic bronchoscopy (ssRAB). It uses a robot with special sensors to guide a thin tube more accurately to lung nodules than current methods.

Who can join? Adults aged 19 or older who have lung nodules that need tissue sampling and are healthy enough for the procedure.

What happens? Participants will have the robotic procedure while asleep under anesthesia. The robot guides a thin tube to the lung nodule to take a small tissue sample. Participants are watched for problems and followed for 6 months.

What are the risks and benefits? The new technology may be more accurate and safer than current methods. The main risks are small chance of lung collapse or bleeding, similar to regular procedures.

Why is this important? This study will show if the new robotic technology works well and is safe in Korea. If successful, it could help diagnose lung cancer earlier and more accurately.

This study will include 100 people at Ulsan University Hospital in Korea.

DETAILED DESCRIPTION:
Background and Rationale:

Peripheral pulmonary nodules (PPNs) are increasingly detected due to widespread use of computed tomography (CT) imaging and lung cancer screening programs. Current bronchoscopic diagnostic methods, including electromagnetic navigation bronchoscopy (ENB) and radial endobronchial ultrasound (rEBUS), have diagnostic yields of approximately 70%, with lower success rates for smaller nodules (<20mm), nodules in the outer third of the lung, and those without bronchus sign.

The ION endoluminal system (Intuitive Surgical, Sunnyvale, CA) represents a novel approach using shape-sensing robotic-assisted bronchoscopy (ssRAB) technology. This system employs shape-sensing fiber optics throughout the catheter length to provide real-time catheter position and orientation monitoring, enabling precise navigation and stable positioning capabilities. International studies have reported diagnostic yields of 87-90% with favorable safety profiles.

Study Design and Methodology:

This is a prospective, single-center, observational cohort study designed to evaluate the diagnostic performance and safety of ssRAB in Korean patients. The study will be conducted as part of routine clinical care, with ssRAB replacing conventional bronchoscopy for eligible patients requiring histological diagnosis of peripheral lung nodules.

Pre-procedure Planning:

All participants will undergo thin-section chest CT (≤1.25mm thickness) for 3D navigation planning using PlanPoint Planning Laptop software. Target nodule characteristics, approach pathways, and procedure strategy will be determined prior to the procedure.

Procedure Protocol:

The ssRAB procedure will be performed under deep sedation or general anesthesia using an 8.0mm or larger endotracheal tube. The procedure involves:

1. Initial airway assessment using conventional flexible bronchoscopy
2. ION system docking to the endotracheal tube
3. Vision probe insertion through the ION catheter (3.5mm outer diameter, 2mm working channel)
4. System registration to align navigation mapping with patient anatomy
5. Catheter navigation to target nodule
6. Vision probe removal and radial EBUS confirmation (when applicable)
7. Tissue sampling using various tools (Flexision biopsy needles, forceps, brush, or cryobiopsy)
8. Fluoroscopic guidance when needed
9. Rapid on-site evaluation (ROSE) when available

Safety Monitoring:

All procedure-related complications will be documented according to CTCAE v5.0 criteria. Post-procedure monitoring includes chest imaging to assess for pneumothorax and clinical observation for bleeding, infection, or other adverse events. Participants will be followed for 24 hours post-procedure for immediate complications.

Follow-up and Diagnosis Confirmation:

Participants will be followed for 6 months to establish final diagnosis. For non-specific benign findings, final diagnosis will be confirmed through additional procedures (surgery or CT-guided biopsy) or 6-month follow-up imaging showing nodule improvement or resolution.

Statistical Analysis:

The primary endpoint is diagnostic yield, defined as the proportion of lesions with definitive diagnosis among total sampled lesions. Secondary endpoints include navigation success rate, rEBUS confirmation rate, procedural performance metrics (registration time, navigation time, total procedure time, fluoroscopy time), and safety outcomes. Based on previous studies reporting 87.8% diagnostic yield, a sample size of 100 patients provides adequate power with 95% confidence interval and ±7% margin of error, accounting for 10% dropout rate.

Expected Impact:

This study will provide the first Korean data on ssRAB performance and safety, potentially establishing evidence for broader implementation of this technology in Korea. The results may contribute to improved diagnostic accuracy for peripheral lung nodules and better patient outcomes through earlier and more accurate diagnosis of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older
* Solid or part-solid peripheral pulmonary nodules confirmed on chest computed tomography (CT)
* Patients requiring histological diagnosis as determined by the treating physician
* Patients eligible for bronchoscopy procedure
* Ability to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 or equivalent functional status allowing procedure under sedation or general anesthesia

Exclusion Criteria:

* Pure ground glass opacity nodules
* Bleeding tendency defined as platelet count less than 50,000/μL or International Normalized Ratio (INR) greater than 1.5
* Severe cardiopulmonary dysfunction precluding deep sedation or general anesthesia
* Pregnant or breastfeeding women
* Life expectancy less than 6 months as assessed by the treating physician
* Inability or unwillingness to provide informed consent
* Absolute contraindication to bronchoscopy including:

  * Severe hypoxemia (oxygen saturation <90% on room air)
  * Severe pulmonary hypertension
  * Recent myocardial infarction (within 6 weeks)
  * Unstable angina
  * Malignant arrhythmias
* Participation in another interventional clinical trial that may interfere with study procedures or outcomes

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with peripheral pulmonary nodules detected on chest CT imaging who require tissue sampling for histological diagnosis. Participants will be recruited from patients referred to the pulmonology department for evaluation of lung nodules. The study population includes patients with solid or part-solid nodules suspicious for malignancy or requiring tissue confirmation for clinical management decisions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield (Proportion of lesions with definitive diagnosis) | At time of procedure and 6 months follow-up
  The proportion of lesions with definitive diagnosis among total biopsied lesions using shape-sensing robotic-assisted bronchoscopy (ssRAB). Diagnostic results are defined as malignant findings, specific benign findings (e.g., tuberculosis, hamartoma), or non-specific benign findings confirmed by additional procedures or 6-month follow-up imaging showing nodule improvement or resolution.

SECONDARY OUTCOMES:
Navigation Success Rate | At time of procedure (Day 0)
  The proportion of successful catheter navigation to target nodules using the ION endoluminal system among all attempted procedures.
Radial EBUS Confirmation Rate | At time of procedure (Day 0)
  The proportion of target nodules confirmed by radial endobronchial ultrasound (rEBUS) among procedures where rEBUS was attempted.
Sensitivity for Malignant Nodules | 6 months follow-up
  The proportion of malignant nodules correctly identified by ssRAB among all nodules confirmed to be malignant by final diagnosis.
Incidence of Procedure-related Complications | 24 hours post-procedure
  Incidence of procedure-related complications including pneumothorax, bleeding (>50mL), infection, and other adverse events. Complications will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Tissue Sample Adequacy (Proportion of procedures yielding adequate tissue samples) | Within 1 week post-procedure
  The proportion of procedures yielding adequate tissue samples for histopathological diagnosis, as determined by the pathologist.
Proportion of procedures with adequate Rapid On-Site Evaluation (ROSE) Results | At time of procedure (Day 0)
  Results of rapid on-site cytological evaluation when performed, including diagnostic adequacy and preliminary findings.

CONTACTS AND LOCATIONS:
Overall Officials: Ganghee Chae, MD, PhD, Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie F, Zhang Q, Mu C, Zhang Q, Yang H, Mao J, Simoff MJ, Huang J, Zhang X, Sun J. Shape-sensing Robotic-assisted Bronchoscopy (SS-RAB) in Sampling Peripheral Pulmonary Nodules: A Prospective, Multicenter Clinical Feasibility Study in China. J Bronchology Interv Pulmonol. 2024 Aug 8;31(4):e0981. doi: 10.1097/LBR.0000000000000981. eCollection 2024 Oct 1. PMID 39115240
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Reisenauer J, Simoff MJ, Pritchett MA, Ost DE, Majid A, Keyes C, Casal RF, Parikh MS, Diaz-Mendoza J, Fernandez-Bussy S, Folch EE. Ion: Technology and Techniques for Shape-sensing Robotic-assisted Bronchoscopy. Ann Thorac Surg. 2022 Jan;113(1):308-315. doi: 10.1016/j.athoracsur.2021.06.086. Epub 2021 Aug 8. PMID 34370981
- [Background] Ost DE, Ernst A, Lei X, Kovitz KL, Benzaquen S, Diaz-Mendoza J, Greenhill S, Toth J, Feller-Kopman D, Puchalski J, Baram D, Karunakara R, Jimenez CA, Filner JJ, Morice RC, Eapen GA, Michaud GC, Estrada-Y-Martin RM, Rafeq S, Grosu HB, Ray C, Gilbert CR, Yarmus LB, Simoff M; AQuIRE Bronchoscopy Registry. Diagnostic Yield and Complications of Bronchoscopy for Peripheral Lung Lesions. Results of the AQuIRE Registry. Am J Respir Crit Care Med. 2016 Jan 1;193(1):68-77. doi: 10.1164/rccm.201507-1332OC. PMID 26367186
- [Background] Nadig TR, Thomas N, Nietert PJ, Lozier J, Tanner NT, Wang Memoli JS, Pastis NJ, Silvestri GA. Guided Bronchoscopy for the Evaluation of Pulmonary Lesions: An Updated Meta-analysis. Chest. 2023 Jun;163(6):1589-1598. doi: 10.1016/j.chest.2022.12.044. Epub 2023 Jan 11. PMID 36640994
- [Background] MacMahon H, Naidich DP, Goo JM, Lee KS, Leung ANC, Mayo JR, Mehta AC, Ohno Y, Powell CA, Prokop M, Rubin GD, Schaefer-Prokop CM, Travis WD, Van Schil PE, Bankier AA. Guidelines for Management of Incidental Pulmonary Nodules Detected on CT Images: From the Fleischner Society 2017. Radiology. 2017 Jul;284(1):228-243. doi: 10.1148/radiol.2017161659. Epub 2017 Feb 23. PMID 28240562
- [Background] Kang MJ, Won YJ, Lee JJ, Jung KW, Kim HJ, Kong HJ, Im JS, Seo HG; Community of Population-Based Regional Cancer Registries. Cancer Statistics in Korea: Incidence, Mortality, Survival, and Prevalence in 2019. Cancer Res Treat. 2022 Apr;54(2):330-344. doi: 10.4143/crt.2022.128. Epub 2022 Mar 16. PMID 35313102
- [Background] Gould MK, Tang T, Liu IL, Lee J, Zheng C, Danforth KN, Kosco AE, Di Fiore JL, Suh DE. Recent Trends in the Identification of Incidental Pulmonary Nodules. Am J Respir Crit Care Med. 2015 Nov 15;192(10):1208-14. doi: 10.1164/rccm.201505-0990OC. PMID 26214244
- [Background] Folch EE, Labarca G, Ospina-Delgado D, Kheir F, Majid A, Khandhar SJ, Mehta HJ, Jantz MA, Fernandez-Bussy S. Sensitivity and Safety of Electromagnetic Navigation Bronchoscopy for Lung Cancer Diagnosis: Systematic Review and Meta-analysis. Chest. 2020 Oct;158(4):1753-1769. doi: 10.1016/j.chest.2020.05.534. Epub 2020 May 23. PMID 32450240
- [Background] Benn BS, Romero AO, Lum M, Krishna G. Robotic-Assisted Navigation Bronchoscopy as a Paradigm Shift in Peripheral Lung Access. Lung. 2021 Apr;199(2):177-186. doi: 10.1007/s00408-021-00421-1. Epub 2021 Feb 6. PMID 33547938
- [Background] Ali MS, Sethi J, Taneja A, Musani A, Maldonado F. Computed Tomography Bronchus Sign and the Diagnostic Yield of Guided Bronchoscopy for Peripheral Pulmonary Lesions. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2018 Aug;15(8):978-987. doi: 10.1513/AnnalsATS.201711-856OC. PMID 29877715